CLINICAL TRIAL: NCT05744609
Title: Development and Validation of a Risk Score for Predicting Severe Outcomes Among Children Hospitalized With Community-acquired Pneumonia
Brief Title: Predicting Severe Outcomes Among Children Hospitalized With Community-acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230203
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Child; Prognosis
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children hospitalized with community-acquired pneumonia
  Interventions: Other: exposures of interest: epidemiological data, clinical characteristics, laboratory data, and chest radiographic reports

INTERVENTIONS:
Other: exposures of interest: epidemiological data, clinical characteristics, laboratory data, and chest radiographic reports — epidemiological data (e.g., age, sex, and residential area), clinical characteristics (e.g., fever, cough, and wheeze), laboratory data (e.g., white blood cell, c-reaction protein, and procalcitonin), and chest radiographic reports (e.g., X-ray, CT, and ultrasound)

SUMMARY:
In this study, investigators aimed to develop and validate a risk score to predict severe outcomes (e.g., mortality and ICU admission) in children who were admitted to the Children's Hospital of Fudan University between 2017 and 2022 due to community-acquired pneumonia (CAP). The objectives were as follows.

1. Develop a risk prediction model based on demographic, comorbidity, clinical characteristics, laboratory data, and chest radiographic reports to predict severe outcomes among children hospitalized with CAP;
2. Develop a risk scoring system and determine the cut-off point;
3. Externally validate the easy-to-use risk score.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 29 days and 18 years old;
2. Admitted to hospital with signs or symptoms of acute infection (eg, fever) and acute respiratory illness (eg, cough), and radiographic evidence of pneumonia.

Exclusion Criteria:

1. Pneumonia developed 48 hours after admission or intubation;
2. Chronic pneumonia, tuberculosis, tracheobronchial foreign bodies, aspiration pneumonia, parasitic lung disease, and diffuse pulmonary interstitial/parenchyma disease.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This was a retrospective cohort study of children aged between > 29 days and 18 years old who were admitted to the Children's Hospital of Fudan University in Shanghai, China from January 1, 2017 to December 31, 2022. Children were enrolled if they were hospitalized with signs and symptoms of lower respiratory tract infection and radiographic evidence of pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | from admission to discharge, an average of 7 days
  in-hospital mortality among children hospitalized with CAP

SECONDARY OUTCOMES:
admission to ICU | from admission to discharge, an average of 7 days
  admission to a intensive care unit for over 24 hours
septic shock | from admission to discharge, an average of 7 days
  occurrence of septic shock during admission
treatment for severe pneumonia | from admission to discharge, an average of 7 days
  vasoactive agents, positive-pressure ventilation or chest drainage, or extracorporeal membrane oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Background] Tseng CC, Tu CY, Chen CH, Wang YT, Chen WC, Fu PK, Chen CM, Lai CC, Kuo LK, Ku SC, Fang WF. Significance of the Modified NUTRIC Score for Predicting Clinical Outcomes in Patients with Severe Community-Acquired Pneumonia. Nutrients. 2021 Dec 31;14(1):198. doi: 10.3390/nu14010198. PMID 35011073
- [Background] Florin TA, Ambroggio L, Brokamp C, Zhang Y, Rattan M, Crotty E, Belsky MA, Krueger S, Epperson TN 4th, Kachelmeyer A, Ruddy R, Shah SS. Biomarkers and Disease Severity in Children With Community-Acquired Pneumonia. Pediatrics. 2020 Jun;145(6):e20193728. doi: 10.1542/peds.2019-3728. Epub 2020 May 13. PMID 32404432
- [Background] Jain S, Williams DJ, Arnold SR, Ampofo K, Bramley AM, Reed C, Stockmann C, Anderson EJ, Grijalva CG, Self WH, Zhu Y, Patel A, Hymas W, Chappell JD, Kaufman RA, Kan JH, Dansie D, Lenny N, Hillyard DR, Haynes LM, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Finelli L; CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. N Engl J Med. 2015 Feb 26;372(9):835-45. doi: 10.1056/NEJMoa1405870. PMID 25714161
- [Background] Florin TA, Ambroggio L, Lorenz D, Kachelmeyer A, Ruddy RM, Kuppermann N, Shah SS. Development and Internal Validation of a Prediction Model to Risk Stratify Children With Suspected Community-Acquired Pneumonia. Clin Infect Dis. 2021 Nov 2;73(9):e2713-e2721. doi: 10.1093/cid/ciaa1690. PMID 33159514